CLINICAL TRIAL: NCT04341454
Title: A Multi-Center, Double-blind, Randomized, Placebo-controlled, Parallel-Group, Phase 3, Therapeutic Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of DWP14012 in Patients With Acute or Chronic Gastritis
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Acute or Chronic Gastritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP14012305
Record Dates: First submitted 2020-04-09; First posted 2020-04-10 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Acute Gastritis; Chronic Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWP14012 X mg QD (Experimental): * Morning: 1 tablet of DWP14012 X mg + 1 tablet of DWP14012 Y mg placebo
  * Evening: 1 tablet of DWP14012 Y mg placebo
  Interventions: Drug: DWP14012 X mg; Drug: DWP14012 Y mg placebo
- DWP14012 Y mg BID (Experimental): * Morning: 1 tablet of DWP14012 X mg placebo + 1 tablet of DWP14012 Y mg
  * Evening: 1 tablet of DWP14012 Y mg
  Interventions: Drug: DWP14012 X mg placebo; Drug: DWP14012 Y mg
- placebo (Placebo Comparator): * Morning: 1 tablet of DWP14012 X mg placebo + 1 tablet of DWP14012 Y mg placebo
  * Evening: 1 tablet of DWP14012 Y mg placebo
  Interventions: Drug: DWP14012 X mg placebo; Drug: DWP14012 Y mg placebo

INTERVENTIONS:
Drug: DWP14012 X mg — DWP14012 X mg, tablet, orally, once daily for 2 weeks
  Arms: DWP14012 X mg QD
Drug: DWP14012 X mg placebo — DWP14012 X mg placebo-matching tablet, orally, once daily for 2 weeks
  Arms: DWP14012 Y mg BID; placebo
Drug: DWP14012 Y mg — DWP14012 Y mg, tablet, orally, twice daily for 2 weeks
  Arms: DWP14012 Y mg BID
Drug: DWP14012 Y mg placebo — DWP14012 Y mg placebo-matching tablet, orally, twice daily for 2 weeks
  Arms: DWP14012 X mg QD; placebo

SUMMARY:
The purpose of study is to confirm the efficacy of DWP14012 X mg QD, DWP14012 Y mg BID compared to placebo in patients with Acute or Chronic Gastritis

DETAILED DESCRIPTION:
This study was designed as a multi-center, randomized, double-blind, placebo-controlled, parallel-group, phase 3 study to assess the efficacy and safety of oral administration of DWP14012 X mg QD, Y mg BID and placebo for 2 weeks in patients with acute and chronic gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 19 and 75 years old based on the date of written agreement
* Those who are diagnosed with acute or chronic gastritis with at least one erosion observed on upper gastrointestinal endoscopy
* Those who had experienced one or more subjective symptoms of gastritis

Exclusion Criteria:

* Those who have had surgery to reduce gastric acid secretion, or gastric or esophageal surgery
* Those with history of clinically significant hepatic, renal, neurologic, pulmonary, endocrine, hematologic, cardiovascular or genitourinary disease that could affect the study results

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Improvement rate of gastric mucosal erosion | at 2 weeks after the IP administration
  Improvement rate (%) = (Number of effective cases(change of ≥ 50% in erosion score) / Number of target cases) x 100

SECONDARY OUTCOMES:
Cure rate of gastric mucosal erosion | at 2 weeks after the IP administration
  Cure rate (%) = (Number of healed cases(0 erosions) / Number of target cases) x 100
Cure rate of gastric mucosal edema | at 2 weeks after the IP administration
  Cure rate (%) = (Number of healed cases(change of 2 to 1 in edema score) / Number of target cases) x 100
Improvement rate of gastric mucosal erythema | at 2 weeks after the IP administration
  Improvement rate (%) = (Number of effective cases(change of ≥ 50% in erythema score) / Number of target cases) x 100
Improvement rate of gastric mucosal bleeding | at 2 weeks after the IP administration
  Improvement rate (%) = (Number of effective cases(change of ≥ 50% in bleeding score) / Number of target cases) x 100
Improvement rate of subjective symptoms | at 2 weeks after the IP administration
  Improvement rate (%) = (Number of effective cases(change of ≥ 50% in subjective symptom score) / Number of target cases) x 100

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim GH, Choi MG, Kim JI, Lee ST, Chun HJ, Lee KL, Choi SC, Jang JY, Lee YC, Kim JG, Kim KB, Shim KN, Sohn CI, Kim SK, Kim SG, Jang JS, Kim N, Jung HY, Park H, Huh KC, Lee KJ, Hong SJ, Baek S, Han JJ, Lee OY. Efficacy and Safety of Fexuprazan in Patients with Acute or Chronic Gastritis. Gut Liver. 2023 Nov 15;17(6):884-893. doi: 10.5009/gnl220457. Epub 2023 Feb 15. PMID 36789577